CLINICAL TRIAL: NCT03800433
Title: Impact of Pentoxifylline Administration on the Modulation of Hyporesponsiveness to Erythropoietin Stimulating Agents in Hemodialysis Patients
Brief Title: Pentoxifylline Administration in Hemodialysis Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Mohamed Elmetwaly, Post grad, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pentoxifylline in hemodialysis
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Anemia Renal
Keywords: pentoxifylline
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): 23 patients will receive their usual dose of erythropoietin stimulating agents and their routine treatment.
- test (Experimental): 23 patients will receive the intervention drug Pentoxifylline (Trental 400 milligram(MG) Extended Release Oral Tablet) twice daily in addition their usual dose of erythropoietin stimulating agents and their routine treatment.
  Interventions: Drug: Trental 400 MG Extended Release Oral Tablet

INTERVENTIONS:
Drug: Trental 400 MG Extended Release Oral Tablet — oral tablets
  Arms: test

SUMMARY:
The aim of the study is to assess the impact of pentoxifylline administration on the modulation of hyporesponsiveness to erythropoietin stimulating agents in hemodialysis patients

DETAILED DESCRIPTION:
this is a prospective, randomized, controlled study to assess the impact of pentoxifylline administration on the modulation of hyporesponsiveness to erythropoietin stimulating agents in hemodialysis patients by determining several outcomes from the intervention and control groups at the end of the study.These outcomes include;the difference in hemoglobin and hematocrit concentration , the difference in inflammatory markers tumor necrosis factor Alpha (TNF-α), interleukin-1 Beta (IL-1β),the difference in the dosage of erythropoiesis stimulating agents ,and The erythropoietin stimulating agents (ESA) resistance index (ERI).

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or over).
* Stable hemodialysis >6 months.
* Regular haemodialysis (3 times/ week).
* ESA resistant anemia (Hb <10 mg/dl for 6 mo.).
* ESA dose of >8000 IU/wk.

Exclusion Criteria:

* Inadequate hemodialysis.
* Hyperparathyroidism (PTH>800 pg/l).
* Known hypersensitivity to, or intolerance of Pentoxifylline.
* Absolute or functional iron deficiency (ferritin < 100 μg/L and/or transferrin saturation < 20%).
* Presence of systemic haematological disease (including antibody-mediated pure red cell aplasia) or known haemoglobinopathy.
* Major surgery, infection, inflammatory diseases, acute myocardial infarction or malignancy within the last 3 months.
* Patients with chronic liver disease and patients who had received immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
The difference in hemoglobin and hematocrit concentration between the intervention and control groups at the end of the study | up to 6 months post baseline
  Patients will be evaluated regularly every month for hemoglobin concentration
safety & tolerability of pentoxifylline ( frequency of adverse drug effects due to Pentoxifylline as well as compliance with pentoxifylline). | up to 6 months post baseline
  Patients will be evaluated regularly for frequency of adverse drug effects due to Pentoxifylline as well as compliance with pentoxifylline

SECONDARY OUTCOMES:
Inflammatory markers TNF-a, IL-1β. | up to 6 months post baseline
  patient will be subjected to laboratory evaluation for estimation of IL-1β,TNF-α levels at baseline as well as end of study evaluation
Difference in the dosage of erythropoiesis stimulating agents. | up to 6 months post baseline
  the dose of ESA will be assessed at end of study evaluation
The ESA ( erythropoiesis stimulating agents)resistance index (ERI). | up to 6 months post baseline
  ERI will be assessed for patients by determining ESA dose and hemoglobin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Lamia El Wakeel, Ass.Prof, Study Director — Ass.prof clinical pharmacy; Radwa El Borolossy, Phd, Study Director — Lecturer of clinical pharmacy; Magdy ElSharkawy, Prof.Dr., Principal Investigator — Prof. of nephrology

REFERENCES:
- [Background] Weiss G, Goodnough LT. Anemia of chronic disease. N Engl J Med. 2005 Mar 10;352(10):1011-23. doi: 10.1056/NEJMra041809. No abstract available. PMID 15758012
- [Background] Johnson DW, Pollock CA, Macdougall IC. Erythropoiesis-stimulating agent hyporesponsiveness. Nephrology (Carlton). 2007 Aug;12(4):321-30. doi: 10.1111/j.1440-1797.2007.00810.x. PMID 17635745
- [Background] Cooper A, Mikhail A, Lethbridge MW, Kemeny DM, Macdougall IC. Pentoxifylline improves hemoglobin levels in patients with erythropoietin-resistant anemia in renal failure. J Am Soc Nephrol. 2004 Jul;15(7):1877-82. doi: 10.1097/01.asn.0000131523.17045.56. PMID 15213276
- [Background] Ferrari P, Mallon D, Trinder D, Olynyk JK. Pentoxifylline improves haemoglobin and interleukin-6 levels in chronic kidney disease. Nephrology (Carlton). 2010 Apr;15(3):344-9. doi: 10.1111/j.1440-1797.2009.01203.x. PMID 20470305
- [Background] Goicoechea M, Garcia de Vinuesa S, Quiroga B, Verdalles U, Barraca D, Yuste C, Panizo N, Verde E, Munoz MA, Luno J. Effects of pentoxifylline on inflammatory parameters in chronic kidney disease patients: a randomized trial. J Nephrol. 2012 Nov-Dec;25(6):969-75. doi: 10.5301/jn.5000077. PMID 22241639
- [Background] Ogawa T, Nitta K. Erythropoiesis-stimulating agent hyporesponsiveness in end-stage renal disease patients. Contrib Nephrol. 2015;185:76-86. doi: 10.1159/000380972. Epub 2015 May 19. PMID 26023017
- [Background] Shahbazian H, Ghorbani A, Zafar-Mohtashami A, Balali A, AleAli A, Lashkarara GR. Administration of pentoxifylline to improve anemia of hemodialysis patients. J Renal Inj Prev. 2016 Nov 26;6(1):61-64. doi: 10.15171/jrip.2017.11. eCollection 2017. PMID 28487874